CLINICAL TRIAL: NCT03464838
Title: The Role of Neuromodulation for Cognitive Processing and Behavioural Inhibition in Gambling Disorder
Brief Title: Effects of Transcranial Direct Current Stimulation (tDCS) in Gambling Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of East London (Other)
Collaborators: GambleAware (Unknown); National Problem Gambling Clinic (Unknown)
Responsible Party: Principal Investigator, Elena Gomis Vicent, Principal Investigator, University of East London
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UREC 1718 23; 241677 (Other: Integrated Research Application System)
Record Dates: First submitted 2018-02-27; First posted 2018-03-14 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Pathological Gambling
MeSH Terms: conditions — Gambling | interventions — Transcranial Direct Current Stimulation; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Investigation of the effects of transcranial direct current stimulation (tDCS) in combination with cognitive behavioural therapy (CBT) against the effects of CBT alone.
Who Masked: Participant, Investigator
Masking Description: Participants will be allocated either to a tDCS Stimulation condition or to a tDCS Sham condition. Neither the investigator nor the participant will know to which condition the participant has been allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real Stimulation tDCS with CBT (Experimental): 16 participants will attend to one weekly tDCS stimulation session with intensity 1.8 milliamps for 8 consecutive weeks. Following the tDCS session, participants will attend to a cognitive behavioural therapy (CBT) session. One tDCS + CBT session per week (Total: 8 sessions).
  Interventions: Device: Transcranial direct current stimulation (tDCS); Behavioral: Cognitive Behavioural Therapy (CBT)
- Sham tDCS with CBT (Sham Comparator): 16 participants will attend to one weekly Sham tDCS session with intensity 0 milliamps for 8 consecutive weeks. Following the Sham tDCS session, participants will attend to a CBT session. One Sham tDCS + CBT session per week (Total: 8 sessions).
  Interventions: Device: Transcranial direct current stimulation (tDCS); Behavioral: Cognitive Behavioural Therapy (CBT)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Transcranial direct current stimulation (tDCS) is a form of noninvasive brain stimulation that applies a very low electrical current to the scalp. tDCS will be applied with intensity of 1.8 milliamps in real stimulation condition and 0 milliamps in sham condition, during 20 minutes, using a high density (HD) tDCS montage over the Prefrontal Cortex (PFC). Electroencephalography (EEG) resting state activity will be measured before and after tDCS.
  Other Names: Noninvasive brain stimulation
Behavioral: Cognitive Behavioural Therapy (CBT) — Cognitive Behavioural Therapy (CBT) is the current treatment available for disordered gamblers at the UK National Problem Gambling Clinic. During the therapy sessions patients acquire learning strategies, cognitive and motivational elements, and develop personal skills to help them improve the understanding of their problems.

SUMMARY:
Gambling disorder is associated to high impulsivity and excessive risk-taking behaviour. These behavioural characteristics related to addiction are linked to cognitive processes in specific brain areas located in the prefrontal cortex (PFC).

With the aim of studying the role of PFC in gambling disorder, the investigators employ transcranial current direct stimulation (tDCS), a noninvasive brain stimulation technique that applies a very weak electrical current to the superficial areas of the brain.

The clinical phase of the research consists on studying the effects of tDCS in combination with cognitive behavioural therapy (CBT) in patients that attend the United Kingdom (UK) National Problem Gambling Clinic. The main objective of the project is to investigate whether the combination of tDCS and CBT can help to decrease impulsivity and risk-taking behaviour and therefore improve the treatment for gambling disorder.

DETAILED DESCRIPTION:
The investigators aim to have a total of 32 participants diagnosed with gambling disorder with the Problem Gambling Severity Index (PGSI). There will be 16 participants per group having two different groups (real stimulation and sham). Real stimulation involves the application of tDCS stimulation and sham condition is used as a control (similar to a placebo).

Participants will attend 8 weekly sessions where they receive tDCS stimulation for 20 minutes, while complete CANTAB cognitive tasks that measure cognitive processes such us control inhibition and risk-taking behaviour. Electroencephalography (EEG) activity will be measured before and after tDCS.

Participants will also complete cognitive questionnaires (Pathological Gambling adapted Yale-Brown Obsessive Compulsive Scale (PG-YBOCS), Gambling Symptom Assessment Scale (G-SAS) and Visual Analogue Scale (VAS) for gambling cravings.

ELIGIBILITY:
Inclusion Criteria:

* Male or females between 18-65 years old diagnosed with disordered gambling based on the Problem Gambling Severity Index (PGSI) who can speak and read English and don't have any of the exclusion criteria.

Exclusion Criteria:

1. History or evidence of chronic or residual neurological disease.
2. A pacemaker or deep brain stimulation.
3. Metal implants in head or neck area (e.g. postoperative clips after intracerebral aneurysm; arterial aneurysm in the vascular system, implantation of an artificial hearing aid).
4. Intracerebral ischemia/history of bleeding.
5. Prior evidence of epileptic seizures, history of epilepsy.
6. History of head injury with loss of consciousness.
7. Any serious medical conditions (disease of the internal organs).
8. Pregnancy or breast-feeding.
9. Negative prescreening from the clinic psychiatrist.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in scores on the Yale-Brown Obsessive Compulsive Scale adapted for Pathological Gambling (PG-YBOCS) | Change from baseline PG-YBOCS scores at week 2, 3, 4, 5, 6, 7 and 8
  It is a 10-item questionnaire that measures the gambling severity. The scores range from 0 to 4 in each question and the total score ranges from 0 to 40. The questions 1 to 5 assess urges and thoughts associated with gambling disorder, and the rest assess the behavioral component of the disorder. The total score will be calculated as well as the separate scores. Gambling severity will be higher with higher PG-YBOCS scores.
Change in scores on the Visual Analogue Scale (VAS) | Change from baseline VAS scores at week 2, 3, 4, 5, 6, 7 and 8
  It is a horizontal line which length is 100 mm where the left side corresponds to the lower scores and the right side to the highest scores (it ranges from 0 to 10). The participant will draw a line where the level best represents their gambling cravings at the current time. The score will be calculated by measuring this line (in millimetres). The gambling cravings will be higher with higher VAS scores.
Change in scores on the Gambling Symptom Assessment Scale (G-SAS) | Change from baseline G-SAS scores at week 8
  It is a 12-item scale to measure gambling symptoms. Each of the 12 questions has a score ranging from 0 to 4 based on the last week. It is useful to measure changes during treatment. The total score ranges from 0 to 48. The symptoms severity will be higher with higher G-SAS scores.
Change in scores on the Cambridge Gambling Task (CGT) | Change from baseline CGT scores at week 8
  Measures of gambling behaviour.

SECONDARY OUTCOMES:
Change in scores on the Information Sampling Task (IST) | Change from baseline IST scores at week 2, 3, 4, 5, 6, 7 and 8
  Measures of impulsivity
Change in scores on the Stop Signal Task (SST) | Change from baseline IST scores at week 2, 3, 4, 5, 6, 7 and 8
  Measures of control inhibition
Change in encephalography (EEG) activity | Change from baseline EEG activity in weeks 1, 2, 3, 4, 5, 6, 7 and 8
  Measures of endogenous oscillatory neural activity

CONTACTS AND LOCATIONS:
Locations (1):
- University of East London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
The participant's data are de-identified (i.e. direct and indirect identifiers have been removed and replaced by a code. The researcher is able to link the code to the original identifiers and isolate the participant to whom the data relates).
  The Data Protection Act (1998), is the primary legislation on data storage. It states that personal data can be kept for as long as it is needed in an anonymised state for the study, after which time it must be destroyed.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT03464838/Prot_SAP_002.pdf